CLINICAL TRIAL: NCT06391749
Title: K-ACCELERATE: A Multi-center Prospective Trial to Evaluate Clinical Utility of Multi Cancer Early Detection Test as a Triage Test for Symptomatic Participants
Brief Title: Clinical Validation of an MCED Test in Symptomatic Populations (K-ACCELERATE)
Acronym: K-ACCELERATE
Status: Enrolling by invitation | Type: Observational
Sponsor: Gene Solutions (Industry)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor
Other Study IDs: 04GS
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cancer Colon; Cancer, Liver; Cancer, Lung; Cancer, Breast; Cancer, Gastric
Keywords: Early cancer detection; Circulating Tumour DNA; Liquid biopsy; Vietnam; symptomatic; triage
MeSH Terms: conditions — Colonic Neoplasms; Liver Neoplasms; Lung Neoplasms; Breast Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected from the participants will be processed and analysed the ctDNA to detect cancer in the early stages and to predict the origin of the tumor.
  The residual blood of this test will be stored in -80 degree of Celcius for further testing to: (i) screen or diagnose cancers; (ii) determine the hosts' genetic factors associated with the risks of cancers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate the diagnostic performance of blood-based SPOT-MAS test in symptomatic individuals, the investigators sought to launch a prospective multicenter study, named K-ACCELERATE. The study aims to recruit 1,000 participants who develop symptoms and signs specific to the top five common cancer types including breast, colorectal, gastric, liver and lung cancer.

Primary objective: Evaluate the performance of the SPOT-MAS test in detecting cancer in symptomatic populations.

Secondary objectives: Evaluate the feasibility of incorporating SPOT-MAS as a triage test into primary care to increase the detection rates of malignant cancer while minimizing unnecessary referrals to invasive procedures.

DETAILED DESCRIPTION:
Participants are recruited and referred to one of the five diagnosis pathways according to the participants' symptoms and signs listed.

Before undertaking imaging tests, 10 ml of blood is collected in Streck tube for SPOT-MAS test.

Participants undertake low-resolution imaging (LRI) tests matching with participants' referral diagnosis pathway. Imaging test results are returned within the same day.

If participants get negative results from both SPOT-MAS and LRI, participants will receive treatment for the symptoms based on the standard treatment scheme at hospitals and be followed up for 12 months to confirm their cancer-free status.

- If participants get a positive result from either SPOT-MAS or LRI, participants will be referred to high-resolution imaging tests (HRI) or tissue biopsy to confirm the presence of tumor.

For those with positive results confirming invasive tumors by HRI or tissue biopsy, patients will undergo treatment. The investigators do not provide financial support for their treatment.

For those with no invasive lesions but having positive SPOT-MAS results, participants will be advised to re-take the SPOT-MAS test after 6 months.

If the 2nd SPOT-MAS test results return positive, participants will be advised to perform whole body CT scan. If participants' scanning results return positive, participants will undergo tissue biopsy and treatment.

If the 2nd SPOT-MAS or whole body CT scan is negative, participants will be followed-up for an additional 6 months by surveying to confirm the cancer-free status.

The enrolment is anticipated to last for approximately 6 months

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above Participants are willing and able to give informed consent for participation in the study
* Participants aged over 18 years
* Individuals presenting symptoms associated witht breast, colorectal, gastric, liver and lung cancer (see below) and being referred for low resolution imaging tests including US breast, chest x-ray, colorectal endoscopy, gastroscopy, US abdomen or relevant diagnostic modalities.
* Symptoms and Signs

  * Breast symptoms: Axillary lump/mass; Breast lump/mass; Breast pain; Nipple discharges; Breast skin change
  * Lung symptoms: Symptoms for more than 3 weeks: Dyspnea (shortness of breath); Chest pain; Cough that does not go away; Hemoptysis (coughing up blood)
  * Colorectal symptoms: Hematochezia (blood in the stool); Diarrhea ≥ 3 weeks; Constipation ≥ 3 weeks; Abdominal pain ≥ 3 weeks
  * Gastric symptoms: Epigastric pain ≥ 3 weeks; Hematemesis (vomiting blood)
  * Liver symptoms: Jaundice (yellowing of the skin and eyes); Right upper quadrant (RUQ) pain; Significant weight loss (≥10% of body weight in previous 6 months)
* Consent to undertake high resolution imaging tests or biopsy upon receiving positive test results from either SPOT-MAS or low-resolution imaging tests

Exclusion Criteria:

* Having a history of invasive cancer diagnosed within the last 5 years
* Having undergone treatment for invasive cancer within the last 5 years
* Having a history of bone marrow transplant or whole blood transfusion within the last 3 months
* Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include both males and females, aged 18 or above, who have no history of cancer. Participants are recruited and referred to diagnostic pathways according to the signs and symptoms. The eligible participants will have to satisfy all of the inclusion and exclusion criteria to be recruited into this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of the SPOT-MAS test to detect cancer in symptomatic individuals | 12 months following enrolment
  Sensitivity, Specificity, Positive predictive value, Negative predictive value of the SPOT-MAS test
Evaluate the ability of the SPOT-MAS test to detect tumor tissue origin | 12 months following enrolment
  accuracy of tumor tissue origin identification

SECONDARY OUTCOMES:
Assess the feasibility of using SPOT-MAS as a triage test to assist in decision-making for follow-up high-resolution imaging or tissue biopsy procedures | 12 months following enrolment
  Positive predictive value, Negative predictive value, Sensitivity and Specificity of the SPOT-MAS test in combination with LRI and HRI tests

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Genetics Institute, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of this study may be requested for publication by journals. Sharing anonymised data with future similar/suitable studies will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organisation than authorized in the study.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Lam DL, Pandharipande PV, Lee JM, Lehman CD, Lee CI. Imaging-based screening: understanding the controversies. AJR Am J Roentgenol. 2014 Nov;203(5):952-6. doi: 10.2214/AJR.14.13049. PMID 25341132
- [Background] Allaby M. Referral of suspected cancers: the NICE approach. Lancet Oncol. 2015 Sep;16(12):1229-30. doi: 10.1016/S1470-2045(15)00279-X. No abstract available. PMID 26431865
- [Background] Boeddinghaus I, Johnson SR. Serial biopsies/fine-needle aspirates and their assessment. Methods Mol Med. 2006;120:29-41. doi: 10.1385/1-59259-969-9:29. PMID 16491590
- [Background] Schrag D, Beer TM, McDonnell CH 3rd, Nadauld L, Dilaveri CA, Reid R, Marinac CR, Chung KC, Lopatin M, Fung ET, Klein EA. Blood-based tests for multicancer early detection (PATHFINDER): a prospective cohort study. Lancet. 2023 Oct 7;402(10409):1251-1260. doi: 10.1016/S0140-6736(23)01700-2. PMID 37805216
- [Background] Nicholson BD, Oke J, Virdee PS, Harris DA, O'Doherty C, Park JE, Hamady Z, Sehgal V, Millar A, Medley L, Tonner S, Vargova M, Engonidou L, Riahi K, Luan Y, Hiom S, Kumar H, Nandani H, Kurtzman KN, Yu LM, Freestone C, Pearson S, Hobbs FR, Perera R, Middleton MR. Multi-cancer early detection test in symptomatic patients referred for cancer investigation in England and Wales (SYMPLIFY): a large-scale, observational cohort study. Lancet Oncol. 2023 Jul;24(7):733-743. doi: 10.1016/S1470-2045(23)00277-2. Epub 2023 Jun 20. PMID 37352875
- [Background] Nguyen VTC, Nguyen TH, Doan NNT, Pham TMQ, Nguyen GTH, Nguyen TD, Tran TTT, Vo DL, Phan TH, Jasmine TX, Nguyen VC, Nguyen HT, Nguyen TV, Nguyen THH, Huynh LAK, Tran TH, Dang QT, Doan TN, Tran AM, Nguyen VH, Nguyen VTA, Ho LMQ, Tran QD, Pham TTT, Ho TD, Nguyen BT, Nguyen TNV, Nguyen TD, Phu DTB, Phan BHH, Vo TL, Nai THT, Tran TT, Truong MH, Tran NC, Le TK, Tran THT, Duong ML, Bach HPT, Kim VV, Pham TA, Tran DH, Le TNA, Pham TVN, Le MT, Vo DH, Tran TMT, Nguyen MN, Van TTV, Nguyen AN, Tran TT, Tran VU, Le MP, Do TT, Phan TV, Nguyen HL, Nguyen DS, Cao VT, Do TT, Truong DK, Tang HS, Giang H, Nguyen HN, Phan MD, Tran LS. Multimodal analysis of methylomics and fragmentomics in plasma cell-free DNA for multi-cancer early detection and localization. Elife. 2023 Oct 11;12:RP89083. doi: 10.7554/eLife.89083. PMID 37819044
- [Background] Nguyen THH, Lu YT, Le VH, Bui VQ, Nguyen LH, Pham NH, Phan TH, Nguyen HT, Tran VS, Bui CV, Vo VK, Nguyen PTN, Dang HHP, Pham VD, Cao VT, Nguyen TD, Nguyen LHD, Phan NM, Nguyen TH, Nguyen VTC, Pham TMQ, Tran VU, Le MP, Vo DH, Tran TMT, Nguyen MN, Nguyen TT, Tieu BL, Nguyen HTP, Truong DYA, Cao CTT, Nguyen VT, Le TLQ, Luong TLA, Doan TKP, Dao TT, Phan CD, Nguyen TX, Pham NT, Nguyen BT, Pham TTT, Le HL, Truong CT, Jasmine TX, Le MC, Phan VB, Truong QB, Tran THL, Huynh MT, Tran TQ, Nguyen ST, Tran V, Tran VK, Nguyen HN, Nguyen DS, Nguyen TQT, Phan TV, Do TT, Truong DK, Tang HS, Phan MD, Giang H, Nguyen HN, Tran LS. Clinical validation of a ctDNA-Based Assay for Multi-Cancer Detection: An Interim Report from a Vietnamese Longitudinal Prospective Cohort Study of 2795 Participants. Cancer Invest. 2023 Feb 6:1-17. doi: 10.1080/07357907.2023.2173773. Online ahead of print. PMID 36719061